CLINICAL TRIAL: NCT07377019
Title: The Efficacy and Safety of Pulsatile Compression Boots in Patients With Acute Decompensated Heart Failure. A Randomized, Controlled Trial.
Brief Title: Efficacy and Safety of Compression Boots in Patients With Acute Decompensated Heart Failure.
Acronym: COMPLEX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Freja Sønder Madsen, Principal investigator, MD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COMPLEX
Record Dates: First submitted 2025-09-12; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Acute Decompensated Heart Failure (ADHF)
Keywords: Acute Decompensated Heart Failure; Heart failure; Compression therapy; Cardiorenal syndrome
MeSH Terms: conditions — Heart Failure; Cardio-Renal Syndrome | interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsatile compression boots (PCB) (Experimental): Receives sessions with PCB (YourBoots, CE approved), as an add on intervention during the entire hospital stay. The PCB intervention will be blinded for the treating clinicians as far as possible in a clinical setting. Furthermore, the study will not interfere with the treating clinician' choice of treatment in general.
  Interventions: Device: Pulsatile Compression Boots (PCB)
- Usual care (No Intervention): Receives either no non-pharmacological treatment or the non-pharmacological treatment chosen by the clinician (e.g. compression bandages), but no compression boots.

INTERVENTIONS:
Device: Pulsatile Compression Boots (PCB) — Each boot has eight chambers that can be inflated to between 30 and 240 mmHg. The first chamber that inflates is at ankle level. When this chamber has achieved the predefined pressure for 17 seconds, the next proximal chamber (chamber two) inflates while the pressure in the distal (ankle) chamber is maintained at constant pressure. This sequence continues until the most proximal chamber at the thigh (chamber eight) has been inflated and has held the maximum pressure for 17 seconds. Thereafter, all the chambers open to release the air, and there is a pause for 30 seconds. The sequence then starts again and continues for 30 minutes. This 30-minute sequence is termed one "session". Pulsatile compression therapy will be applied three sessions per day.
  Other Names: Pneumatic compression boots; Intermittent pneumatic compression boots; Sequential compression boots; Pneumatic compression devices; Dynamic compression boots; Pulsatile compression therapy
  Arms: Pulsatile compression boots (PCB)

SUMMARY:
The aim of this clinical trial is to investigate whether pulsatile compression therapy can support heart and kidney function in patients admitted with acute heart failure and fluid accumulation in the legs.

Pulsatile compression boots, which provide pulsatile compression therapy, work by adding a predefined pressure to the legs in a rhythm that enhances mobilization of peripheral edema and improves venous and lymphatic drainage from the lower extremities. This increased venous return (preload) may allow the heart to fill more effectively and pump more strongly, thereby improving circulation. Better circulation can enhance kidney blood flow, help diuretics work more efficiently, and reduce the risk of complications due to worsening heart failure, affecting both the heart and kidneys.

The investigators want to explore whether adding this therapy to standard diuretic treatment is safe, feasible, and offers benefits compared with standard diuretic treatment alone.

Participants will receive three daily sessions of pulsatile compression therapy alongside usual clinical care.

DETAILED DESCRIPTION:
Background:

Compression therapy is an effective treatment for fluid accumulation in the legs (leg edema). Nevertheless, it is only used sporadically and inconsistently in patients with acute heart failure (HF) and leg edema, even though leg edema is a major problem in these hospitalized patients and compression therapy could help alleviate it.

Acute HF is often complicated by leg edema, which causes pain, reduced mobility, and consequently reduced quality of life. It is well-known that compression therapy can reduce leg edema and is standard treatment for leg edema caused by venous and lymphatic disease, but not for HF. Currently, the standard treatment for HF-related leg edema is diuretic medication. However, this is associated with challenges such as worsening kidney function and prolonged hospitalizations.

No randomized controlled trials have evaluated compression therapy as an adjunct to diuretics in HF, and neither Danish nor European HF guidelines mention its use. This represents an important knowledge gap.

Pulsatile compression therapy are a relatively new modality that mimic the natural muscular venous pump activated during walking. Studies show that compression therapy can increase venous return to the heart. This may potentially improve cardiac function, according to the Frank-Starling mechanism, and enhance renal blood flow, thereby allowing more effective fluid removal.

Pulsatile compression therapy thus represents a non-pharmacological approach with the potential to reduce edema, optimize decongestion, shorten hospitalization, and improve quality of life in this large patient population.

This project investigates the clinical efficacy and safety of pulsatile compression therapy in patients hospitalized with acute HF and leg edema through a randomized controlled trial, which will provide important clinical knowledge on compression therapy for HF patients

Aim:

This randomized, controlled clinical trial will evaluate the efficacy, safety, and feasibility of using pulsatile compression therapy in combination with IV diuretics in patients with mild to moderate HF admitted with worsening symptoms and bilateral leg edema. The study is designed to:

1. Assess the impact of pulsatile compression therapy on systolic pulmonary arterial pressure (sPAP), as a key hemodynamic parameter.

Hypothesis:

The investigators hypothesize that treatment with a combination of pulsatile compression therapy and diuretics is a safe and feasible approach. The investigators hypothesize that this combined therapy will safely improve hemodynamic parameters, through the activation of the Frank-Starling mechanism, and subsequently improve renal perfusion, compared with standard diuretic therapy alone. This may optimize diuretic response and reduce the risk of developing cardiorenal syndrome.

Methods:

The COMPLEX study is a prospective, randomized, controlled trial conducted at the Cardiovascular Research Unit in Svendborg Hospital, Denmark. The study population consist of patients hospitalized with acute decompensated HF and bilateral leg edema, who are initiated with intravenous diuretics. Onehundred-and-ten participants are anticipated to take part in the study including a pilot study of 10 participants. Participants are randomized in a 1:1 ratio to receive either treatment with pulsatile compression therapy during hospitalisation, or standard treatment without pulsatile compression therapy. All participants will undergo the following examinations at baseline:

* Ultrasound examination of the heart (echocardiography), the kidneys and the lungs
* Physical examination, including measurement of leg circumference
* Blood- and urine samples
* Registration of "Congestions Score" and "NYHA classification".
* Patient-reported quality of life will be measured using the validated LYMQOL Leg questionnaire.

These examinations will be repeated after the 5th treatment with pulsatile compression therapy (the control group will undergo assessments at a corresponding time point) and at discharge.

Ninety days after discharge, the investigators will review medical records to assess whether participants have experienced a heart failure-related readmission.

Sample size estimation:

A reduction in the primary endpoint of 15% is anticipated in participants assessed in the COMPLEX study compared to usual care. With a power of 0,80 and a two-sided alpha value of 0,05, 90 participants are needed. Accounting for a 10% dropout rate, approximately 100 participants will need to be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving written informed consent
* Inclusion within 24 hours from admission
* Bilateral LE edema - defined as: Pitting edema scale > 1, bilaterally
* Initial IV diuretic treatment

Evidence of heart failure - at least one of the following:

1. Heart failure with reduced ejection fraction (HFrEF):

   * Signs and/or symptoms of HF
   * Left ventricular ejection fraction (LVEF) ≤ 40%
2. Heart failure with mildly reduced ejection fraction (HFmrEF):

   * Signs and/or symptoms of HF
   * LVEF 41 - 49%
3. Heart failure with preserved ejection fraction (HFpEF):

   * Signs and/or symptoms of HF
   * LVEF ≥ 50 %
   * Evidence of structural heart disease (Left atrial enlargement or left ventricular hypertrophy)
   * NT-proBNP > 300pg/mL for patients without ongoing atrial fibrillation/flutter, and NT-proBNP > 600 pg/mL for patients with ongoing atrial fibrillation/flutter.

Evidence of elevated pulmonary artery pressure - at least one of the following:

* Systolic pulmonary artery pressure (sPAP) > 35 mmHg
* Tricuspid regurgitation gradient (TRG) > 30 mmHg
* Severe tricuspid regurgitation and VCI > 20 mm.

Additional echocardiographic criteria:

- Left atrial end-systolic volume index > 34 mL/m2

Exclusion Criteria:

* Pregnancy
* Life expectancy less than 1 year for any reason
* Expected hospital stay less than 1 day
* New York Heart Association classification (NYHA) class IV
* LVEF < 20%
* Diastolic left ventricular diameter > 70 mm
* Known history or symptoms of peripheral arterial disease (Intermittent claudication or brachial-ankle index with value < 0,9)
* Significant leg wounds or infections
* Deep venous thrombosis (DVT)
* Need for treatment with inotropes or vasopressors
* Permanent dialysis
* Manifest acute kidney injury with oliguria
* Current high-pressure pulmonary edema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Change in systolic pulmonary arterial pressure (sPAP) from baseline to hospital discharge. | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by transthoracic echocardiography. sPAP will be used as a surrogate marker of the degree of cardiac backward failure.
  Unit: mmHg

SECONDARY OUTCOMES:
Change in estimated glomerular filtration rate (eGFR) from baseline to hospital discharge. | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by a blood sample. Renal function will be assessed by eGFR, calculated from serum cystatin C, serving as a surrogate marker of renal function Unit: mL/min/1,73m^2
Change in NT-proBNP | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Collected by a blood sample. Unit: ng/L
Change in E/A-ratio | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by transthoracic echocardiography.
  Unit: dimensionless
Change in E/é (septal and lateral) | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by transthoracic echocardiography
  Unit: dimensionless
Change in é septal and lateral | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by transthoracic echocardiography Unit: cm/s
Change in left ventricular ejection fraction (LVEF) | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by transthoracic echocardiography using Simpson's biplane method. Unit: %
Change in Global Longitudinal Strain (GLS) | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by transthoracic echocardiography. Unit: %
Change in left ventricular stroke index | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by transthoracic echocardiography Unit: ml/m^2
Change in cardiac ouput | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by transthoracic echocardiography. Unit: l/min
Change in cardiac index | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by transthoracic echocardiography. Unit: l/min/m^2
Change in left atrial end-systolic volume | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by transthoracic echocardiography using the apical four-chamber view at end-ventricular systole.
  Unit: ml
Change in left atrial end-systolic volume index | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by transthoracic echocardiography using the apical four-chamber view at end-ventricular systole.
  Unit: ml/m^2
Change in left atrial strain | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by transthoracic echocardiography. Unit: %
Change in Tricuspid Annular Plane Systolic Excursion (TAPSE) | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by echocardiography, using M-mode. Unit: mm.
Change in right ventricular s' | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by transthoracic echocardiography. Unit: m/s
Change in right ventricular strain | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by transthoracic echocardiography. Unit: %
Change in right ventricular end-systolic volume index | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by transthoracic 3D echocardiography . Unit: ml/m^2
Change in Right Ventricular end-diastolic volume index | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by transthoracic 3D echocardiography Unit: ml/m^2
Change in right ventricular stroke volume index | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by transthoracic 3D echocardiography Unit: ml/m^2
Change in the diameter of Vena Cava Inferior | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by transthoracic echocardiography. Unit: mm.
Change in renal artery peak systolic velocity | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by ultrasound of the distal segment of the renal artery using pulsed-wave Doppler.
  Unit: cm/s
Change in renal artery end-diastolic velocity | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by ultrasound of the distal segment of the renal artery using pulsed-wave Doppler.
  Unit: cm/s
Change in renal artery resistive index | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by ultrasound of the distal segment of the renal artery using pulsed-wave Doppler.
  Unit: Dimensionless
Change in the time-averaged mean and maximum velocities in the renal artery. | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by ultrasound of the distal segment of the renal artery using pulsed-wave Doppler.
  Unit: cm/s
Change in urine albumin-to-creatinine ratio (UACR) | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by urine sample. Unit: mg/g

OTHER OUTCOMES:
Change in length of hospital stay | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured in hours
Change in pulmonary congestion, assessed by semi-quantitative B-line scoring | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured by focused lung ultrasound examination using a 14-zone protocol. Quantification of B-lines will be performed as a semi-quantitative assessment of pulmonary congestion. B-lines represent increased extravascular lung fluid and are used as a marker of pulmonary congestion.
Change in 30- and 90-day readmission rates | From baseline (Day 1, hospital admission) to 30 and 90 days after discharge
  Readmissions should be related to heart failure
Change in Quality of Life, using LYMQOL-leg questionnaire | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  LYMQOL-leg is a questionnaire designed to measure quality of life in patients with chronic bilateral leg edema or lymphedema.
Change in the dose of intravenous and oral diuretic treatment | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Unit: mg.
Change in daily dosing frequency of intravenous and oral diuretics | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Unit: administration per day
Change in number of days receiving intravenous diuretic therapy. | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  The total number of calendar days during which the patient receives at least one dose of intravenous loop diuretics during the index hospital admission will be recorded. The outcome is defined as the difference in number of days with intravenous diuretic treatment between treatment groups.
  Unit: days
Change in leg circumference | Measured at baseline (Day 1, hospital admission) and at hospital discharge (assessed up to 14 days after admission)
  Measured in millimeter (mm.) at the ankle, calf and thigh.

CONTACTS AND LOCATIONS:
Overall Officials: Freja S. Madsen, M.D., Ph.D student, Principal Investigator — Cardiovascular Research Unit, OUH, Svendborg
Locations (1):
- Cardiovascular Research Unit. Odense University Hospital, Svendborg., Svendborg, Denmark